CLINICAL TRIAL: NCT03416959
Title: Prospective Bone Metastases Database
Brief Title: Bone Metastases Database of Patients Treated Surgically for Impending or Pathologic Fracture of Long Bones
Acronym: BMD
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, MD, PhD., Istituto Ortopedico Rizzoli
Other Study IDs: 0012807
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: intramedullary fixation or endoprosthetic reconstruction — Surgical treatment for long bone metastases with intramedullary nail or endoprosthetic reconstruction

SUMMARY:
The aims of this study are to collect prospective data on the natural history of bone metastases (BMs) and skeleta related events (SREs),

DETAILED DESCRIPTION:
The aims of this study are to evaluate clinical and biological factors of patients with BMs after reconstruction with intramedullary fixation (IMN) or endoprosthetic reconstruction (EPR) with a specific focus on (1) the rate of complication or failure; (2) differences in complication rates by anatomic site; (3) functional results as assessed by the Musculoskeletal Tumor Society System (MSTS); (4) differences in complication rate between patients treated with INM versus EPR; and (5) differences in survival in patients with metastatic bone disease based on disease-specific, laboratory, and demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long bone metastases treated surgically with intramedullary nail or endoprosthetic reconstruction

Exclusion Criteria:

* Patients with bone metastases of the spine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bone metastases in the extremities treated with intramedullary fixation or endoprosthetic recosntruction for impending fracture or pathologic fracture
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes after treatment of long bone metastases with intramedullary nail versus endoprosthetic reconstruction | 24 months
  The study includes the collection of clinical data (age, sex, Karnofsky score) and laboratory data related to the patient (erythrocyte sedimentation rate, C reactive protein, Alkaline phosphatase, white blood cells and hemoglobin) at the time of admission, data on the pathology (histotype, site of bone metastasis , presence of further skeletal or visceral metastases), type of surgery performed (stabilization versus resection).The objectives of this study is to examine clinical outcomes after after surgical treatment of bone metastases with a specific focus on differences in complication rate between patients treated with intramedullary nail versus endoprosthetic reconstruction

SECONDARY OUTCOMES:
Survival in patients undergoing surgery for metastatic bone disease | 24 months
  Provide a reliable and objective means of estimating survival in patients with metastatic bone disease based on disease-specific and laboratory tests

OTHER OUTCOMES:
Prognostic factor regarding erythrocyte sedimentation rate | 24 months
  erythrocyte sedimentation rate (mm/h)
Prognostic factor regarding C reactive protein | 24 months
  C reactive protein (mg/dl)
Prognostic factor regarding Alkaline phosphatase | 24 months
  Alkaline phosphatase (U/L)
Prognostic factor regarding white blood cells | 24 months
  white blood cells (10/mm)
Prognostic factor regarding hemoglobin | 24 months
  hemoglobin (g/dl)
Prognostic factor regarding Karnofsky score | 24 months
  Karnofsky score (0/100)

CONTACTS AND LOCATIONS:
Overall Officials: Costantino Errani, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
The data will be published in the international literature at the end of the study